CLINICAL TRIAL: NCT03621969
Title: Technology Development for Physical Rehabilitation of Patients With Upper Extremity Motor Deficits
Brief Title: Technology Development for Physical Rehabilitation of Patients With Upper Extremity Motor Deficits (RePlay)
Acronym: RePlay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Robert Rennaker, Professor, The University of Texas at Dallas
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 16-74
Record Dates: First submitted 2017-01-25; First posted 2018-08-09 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Spinal Cord Injuries
Keywords: Vagus Nerve Stimulation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Restraint, Physical; Health Records, Personal; Physical Examination

STUDY DESIGN:
Intervention Model Description: Group 1 will receive:
  1. two weeks of RePlay device therapy twice per week at REACT (weeks 1-2), followed by re-assessment,
  2. then will rest for 2 weeks (weeks 3-4),
  3. then will take the RePlay devices and tablet computer home for two weeks (weeks 5-6) for daily device therapy, followed by re-assessment.
  Group 2 will receive:
  1. two weeks of RePlay device therapy daily at home (they will take the devices and tablet home) (weeks 1-2), followed by re-assessment,
  2. then will rest for 2 weeks (weeks 3-4),
  3. then will receive two weeks of RePlay device therapy twice per week at REACT (weeks 5-6), and then will undergo re-assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1 will receive:
  1. Medical History and Brief Physical Exam
  2. Diagnostic Assessments
  3. Patient Instruction and use of RePlay Device
  4. two weeks of RePlay device therapy twice per week at REACT (weeks 1-2), followed by re-assessment,
  5. then will rest for 2 weeks (weeks 3-4),
  6. then will take the RePlay devices and tablets home for two weeks (weeks 5-6) for daily RePlay device therapy, followed by re-assessment.
  Interventions: Other: Physical exam and medical history; Diagnostic Test: Assessments; Device: Patient Instruction and use of Device (RePlay)
- Group 2 (Experimental): Group 2 will receive:
  1. Medical History and Brief Physical Exam
  2. Diagnostic Assessments
  3. Patient Instruction and use of RePlay Device
  4. two weeks of RePlay device therapy daily at home (they will take the RePlay devices and tablets home) (weeks 1-2), followed by re-assessment,
  5. then will rest for 2 weeks (weeks 3-4),
  6. then will receive two weeks of RePlay device therapy twice per week at REACT (weeks 5-6), and then will undergo re-assessment.
  Interventions: Other: Physical exam and medical history; Diagnostic Test: Assessments; Device: Patient Instruction and use of Device (RePlay)

INTERVENTIONS:
Other: Physical exam and medical history — This will be completed by a medical doctor on the research team
Diagnostic Test: Assessments — One assessment in Phase I, and three assessments in Phase II (baseline, and following each 2 week active study period)
Device: Patient Instruction and use of Device (RePlay) — 1. providing measurable upper extremity movement, control, and coordination feedback for patients, therapists, and physicians
  2. improving assessment and evaluation of patients involved in future interventional studies,
  3. producing a dynamic, responsive, inexpensive physical therapy system that can be used in the comfort of the participants' own home.

SUMMARY:
Injuries and disease processes that produce upper extremity deficits are devastating to patients and their families. One potential avenue to treat these neurological disorders is through the enhancement of neural plasticity, which is the ability of the brain to reorganize and recover following insult. After a minor injury, the brain undergoes beneficial neural plasticity, compensating for altered neural activity to restore normal function. However, in the cases of moderate to severe injury and disease, e.g. spinal cord injury (SCI), insufficient or improper plasticity limits recovery, leaving patients with long-term disability. Therefore, methods that can drive robust and specific plasticity have great potential to treat neurological injuries and disease.

The Texas Biomedical Device Center (TXBDC) at UT Dallas has developed a groundbreaking therapy, called Targeted Plasticity Therapy (TPT), which pairs traditional motor, sensory, and cognitive rehabilitation with precise stimulation of the vagus nerve, to guide such robust and specific plasticity to treat a wide range of neurological deficits.

DETAILED DESCRIPTION:
The groundbreaking therapy developed at Texas Biomedical Device Center (TXBDC) , called Targeted Plasticity Therapy (TPT) pairs traditional motor, sensory, and cognitive rehabilitation with precise stimulation of the vagus nerve, to guide such robust and specific plasticity to treat a wide range of neurological deficits. The success of this concomitant therapy will be furthered, in part, through the development and use of mechanical devices aimed at measuring the effects of rehabilitation in patients with an upper extremity neurological deficit, e.g. from SCI. These devices are small hand controllers used to play simple video games that can also measure force and movement. Additionally, this study will be used to inform the future development of the rehabilitation game software as well as an optional game chair (in patients that use wheelchairs, the games can also be played from the patient's own chair).

To optimize the evaluation of these RePlay devices and software, and to decrease the time requirement for patients, research will be divided into two phases. Patients can participate in either one or both phases. Participation in phase II is not contingent on participation in phase I.

Phase I will involve 80 participants using the RePlay devices and games on a single visit. These 80 participants will be a collection of participants with no neurological disorders, participants recovering from stroke, those with Multiple Sclerosis, Parkinson's Disease and Spinal Cord Injuries. This will allow us to determine the ability of these patient populations to enjoyably use these devices and games compared with their degree of impairment. Participants' degree of impairment will be quantified by standard rehabilitation measurements for each disease process, including the ASIA Spinal Cord Impairment Scale, GRASSP, Jebsen Taylor Hand Function, dynomometry strength readings

In Phase II, 20 participants will be randomized equally to one of two groups. Each group will receive the same amount of therapy, only in a different sequence.

Group 1 will receive:

1. two weeks of RePlay device therapy twice per week at REACT (weeks 1-2), followed by re-assessment,
2. then will rest for 2 weeks (weeks 3-4),
3. then will take the RePlay devices and tablets home for two weeks (weeks 5-6) for daily RePlay device therapy, followed by re-assessment.

Group 2 will receive:

1. two weeks of RePlay device therapy daily at home (they will take the devices and tablets home) (weeks 1-2), followed by re-assessment,
2. then will rest for 2 weeks (weeks 3-4),
3. then will receive two weeks of RePlay device therapy twice per week at REACT (weeks 5-6), and then will undergo re-assessment.

This will allow investigators to test the Replay rehabilitation software and hardware over 2 two week periods in order to evaluate the pattern of game play improvement in this population over time in different settings.

ELIGIBILITY:
Inclusion Criteria:

* Partial upper limb impairment in one or both arms as a result of a neurological injury or disease
* Age 18-65

Exclusion Criteria:

* Emotional disability that would interfere with participation as determined by Dr.

Wigginton

* Inability to understand instructions in English
* No upper limb movement
* Incarcerated individuals
* For Phase II, anticipated inability to complete study visits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the rehabilitation device design as reported by subjects using a 10-point Likert scale | Through Study Completion, approximately 8-9 weeks
  Assess feasibility, ease of use and enjoyment for device in injured population. This will be measured by subject report. Subjects will verbally provide feedback as they use the software and hardware. Feedback will be recorded and changes will be made based on feedback received from participants. Subjects self-report their experienced enjoyment of RePlay using a 10-point Likert scale (10 = extreme enjoyment, 1 = no enjoyment). Higher scores represent a greater degree of experienced enjoyment.
Evaluate the functionality of rehabilitation device as reported by subjects using a 10-point Likert scale | Through Study Completion approximately 8-9 weeks
  Assess general fit, and functionality of these devices to further the device development. both in the home and in the rehabilitation setting. This will be measured by subject report. This will be measured by subject report. Subjects will verbally provide feedback as they use the software and hardware. Feedback will be recorded and changes will be made based on feedback received from participants. Subjects self-report their experienced fit and function of RePlay using a 10-point Likert scale (10 = extremely easy to fit, 1 = didn't fit at all). Higher scores represent a greater degree of experienced fit and function

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - REACT, Addison, Texas
  - UT Dallas, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No